CLINICAL TRIAL: NCT05980416
Title: A Phase 1 Dose Escalation and Expansion Study of EO-3021, an Anti-claudin 18.2 (CLDN18.2) Antibody Drug Conjugate, in Patients With Solid Tumors Likely to Express CLDN18.2
Brief Title: Study of EO-3021 in Adult Patients With Solid Tumors Likely to Express CLDN18.2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Elevation Oncology (Industry)
Collaborators: Eli Lilly and Company (Industry); GlaxoSmithKline (Industry); CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELVCAP-002-01
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Stomach Neoplasm; Gastrointestinal Neoplasms; Digestive System Neoplasm; Neoplasms by Site; Neoplasms
Keywords: Gastric Cancer; Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Adenocarcinoma | interventions — Ramucirumab; dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EO-3021 Monotherapy (Experimental): In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma will receive EO-3021 monotherapy at various doses every 3 weeks to determine MTD/RP2D(s).
  In expansion, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma expressing CLDN18.2 who have received one and no more than three lines of prior systemic therapy in the advanced metastatic setting will be randomized to one of two doses of EO-3021 dosed every 3 weeks to confirm RP2D.
  Interventions: Drug: EO-3021
- EO-3021 in combination with ramucirumab (Experimental): In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma will receive EO-3021 at various doses in combination with ramucirumab every 3 weeks to determine MTD/RP2D(s).
  In expansion, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma expressing CLDN18.2 who have received only one prior systemic therapy in the advanced metastatic setting will be treated with EO-3021 in combination with ramucirumab every 3 weeks to confirm RP2D.
  Interventions: Drug: EO-3021; Drug: Ramucirumab (CYRAMZA®)
- EO-3021 in combination with dostarlimab (Experimental): In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma will receive EO-3021 at various doses in combination with dostarlimab every 3 weeks to determine MTD/RP2D(s).
  In expansion, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma expressing CLDN18.2 who have not received any prior systemic therapies in the advanced metastatic setting will be treated with EO-3021 in combination with dostarlimab every 3 weeks to confirm RP2D.
  Interventions: Drug: EO-3021; Drug: Dostarlimab

INTERVENTIONS:
Drug: EO-3021 — Anti-Claudin 18.2 antibody drug conjugate
Drug: Ramucirumab (CYRAMZA®) — VEGFR2 inhibitor
  Arms: EO-3021 in combination with ramucirumab
Drug: Dostarlimab — anti-PD-1 antibody
  Arms: EO-3021 in combination with dostarlimab

SUMMARY:
This study is an open-label, international, multi-center, Phase 1 study in adult patients with solid tumors likely to express CLDN18.2.

ELIGIBILITY:
Key Inclusion Criteria:

* Availability of tumor tissue for evaluation of biomarker
* Patients enrolled to expansion must have tumors expressing CLDN 18.2 based on central prospective IHC testing.
* Histologically and/or cytologically confirmed diagnosis of advanced metastatic gastric/GEJ adenocarcinoma not amenable to resection or radiation therapy with curative intent

  •≥ 18 years of age
* ECOG performance status (PS) 0 or 1 at Screening
* Progressed on or after standard therapy, or are intolerable of available standard therapy, or there is no available standard therapy
* In dose escalation, there is no limit on the number of prior lines of therapy.
* In expansion, for EO-3021 monotherapy, at least 1 but no more than 3 prior lines of therapy in the advanced/metastatic setting is allowed
* In expansion, for EO-3021 in combination with ramucirumab, only 1 prior line of therapy in the advanced/metastatic setting is allowed. Prior fluoropyrimidine and platinum-containing chemotherapy is required
* In expansion, for EO-3021 in combination with dostarlimab, no prior systemic therapy in the advanced/metastatic setting is allowed.
* Have at least one measurable extra-cranial lesion as defined by RECIST v1.1
* Adequate organ function
* Life expectancy > 12 weeks
* Ability to understand the nature of this study, comply with protocol requirements, and give written informed consent
* Willingness of men and women of reproductive potential to observe conventional and effective birth control for the duration of treatment and for 6 months following study completion (or longer if required by local regulation)

Key Exclusion Criteria:

* Pregnant or breastfeeding
* Symptomatic or untreated brain metastases
* Have previously received CLDN18.2 antibody drug conjugates (ADCs) or any ADC containing an auristatin payload (prior monoclonal antibody against CLDN18.2 may be eligible)
* Have peripheral neuropathy Grade ≥2
* Have history of non-infectious pneumonitis/interstitial lung disease
* Have diagnosis of another malignancy, or history of systemic treatment for invasive cancer within last 3 years. Note: Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. Diagnosis of non-melanoma skin cancer, carcinoma in situ of the cervix or breast, or noninvasive tumor does not affect eligibility
* Have active ocular surface disease at baseline (based on screening ophthalmic examination) as defined as symptomatic or Grade ≥2 disease involving the cornea
* Have history of Grade ≥2 gastritis
* Have serious concurrent illness or clinically relevant active bacterial, fungal or viral infection
* Have a history of several allergic and/or anaphylactic reactions to known chimeric, human, or humanized antibodies, fusion proteins or known allergies to components of EO-3021, ramucirumab, or dostarlimab
* Clinically significant cardiac disease, including but not limited to symptomatic congestive heart failure, unstable angina, acute myocardial infarction within 6 months of planned first dose, or unstable cardiac arrhythmia requiring therapy (including torsades de pointes)
* Have history of allogenic hematopoietic stem cell transplantation or solid organ transplantation with ongoing systemic immunosuppressive therapy
* Received any live vaccine within 30 days of enrollment
* Patients who are not appropriate candidates for participation in this clinical study for any other reason as deemed by the Investigator
* Expansion only: Have HER2+ disease as defined by American Society of Clinical Oncology-College of American Pathologists guidelines for gastric/GEJ adenocarcinoma
* Ramucirumab Arms Only: Received prior treatment with ramucirumab and other VEGFR2 inhibitors
* Dostarlimab Arms Only: Prior treatment with immune checkpoint inhibitors (ICI) including dostarlimab and other anti-PD-1, anti-PD-L1, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (16):
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Yale - Smilow Cancer Hospital, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Johns Hopkins University - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Henry Ford Cancer, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health/Wake Forest University, Charlotte, North Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - UW Carbone Cancer Center - Cancer Connect, Madison, Wisconsin
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo Ku, Tokyo
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Yonsei University, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EO-3021 Monotherapy 1.0 mg/kg: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma received EO-3021 monotherapy 1.0 mg/kg every 3 weeks to determine MTD/RP2D(s).
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
- EO-3021 Monotherapy 2.0 mg/kg: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma received EO-3021 monotherapy 2.0 mg/kg every 3 weeks to determine MTD/RP2D(s).
  In expansion, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma expressing CLDN18.2 who had received at least 1 but no more than 3 prior lines of therapy in the advanced metastatic setting were randomized to EO-3021 2.0 mg/kg or 2.5 mg/kg every 3 weeks in a 1:1 fashion.
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
- EO-3021 Monotherapy 2.5 mg/kg: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma received EO-3021 monotherapy 2.5 mg/kg every 3 weeks to determine MTD/RP2D(s).
  In expansion, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma expressing CLDN18.2 who had received at least 1 but no more than 3 prior lines of therapy in the advanced metastatic setting were randomized to EO-3021 2.0 mg/kg or 2.5 mg/kg every 3 weeks in a 1:1 fashion.
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
- EO-3021 Monotherapy 2.9 mg/kg: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma received EO-3021 monotherapy 2.9 mg/kg every 3 weeks to determine MTD/RP2D(s).
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
- EO-3021 2.0 mg/kg in Combination With Ramucirumab: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma received EO-3021 2.0 mg/kg in combination with ramucirumab every 3 weeks to determine MTD/RP2D(s).
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
  Ramucirumab (CYRAMZA®): VEGFR2 inhibitor
- EO-3021 2.0 mg/kg in Combination With Dostarlimab: In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma will receive EO-3021 2.0 mg/kg in combination with dostarlimab every 3 weeks to determine MTD/RP2D(s).
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
  Dostarlimab: anti-PD-1 antibody
Period: Overall Study
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Started | 3 | 42 | 34 | 6 | 2 | 1
Completed | 3 | 42 | 34 | 6 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab | Total
Number analyzed (Participants) | 3 | 42 | 34 | 6 | 2 | 1 | 88
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 67.3 [55.0 to 74.0] | 60.8 [31.0 to 81.0] | 60.7 [31.0 to 82.0] | 65.7 [31.0 to 82.0] | 46.0 [38.0 to 54.0] | 45. [45.0 to 45.0] | 60.8 [31.0 to 83.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2.0 | 15.0 | 8.0 | 1.0 | 1.0 | 1.0 | 28
  Male | 1.0 | 27.0 | 26.0 | 5.0 | 1.0 | 0.0 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0
  Asian | 0.0 | 17.0 | 16.0 | 3.0 | 0.0 | 0.0 | 36
  Native Hawaiian or Other Pacific Islander | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0
  Black or African American | 0.0 | 2.0 | 1.0 | 0.0 | 0.0 | 0.0 | 3
  White | 3.0 | 20.0 | 15.0 | 3.0 | 2.0 | 1.0 | 44
  More than one race | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0
  Unknown or Not Reported | 0.0 | 3.0 | 2.0 | 0.0 | 0.0 | 0.0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events When Treated With EO-3021 as Monotherapy and in Combination With Ramucirumab or Dostarlimab.
Time Frame: From the time of informed consent, for approximately 12 months (or earlier if the participant discontinues from the study), and through Safety Follow-up (28 days after the last dose)
Measure: Count of Participants; unit: Participants
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0
Participants | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0

2. Primary Outcome: The Incidence Rate of Dose Limiting Toxicities (DLT) During the First 21-day Cycle of Treatment With EO-3021 as Monotherapy and in Combination With Ramucirumab or Dostarlimab.
Time Frame: The first 21-day treatment cycle for each patient enrolled in the Escalation Phase
Measure: Count of Participants; unit: Participants
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0
Participants | 0.0 | 0.0 | 2.0 | 5.0 | 0.0 | 0.0

3. Primary Outcome: Number of Patients With Serious Adverse Events When Treated With EO-3021 as Monotherapy and in Combination With Ramucirumab or Dostarlimab.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0
Participants | 2.0 | 20.0 | 15.0 | 4.0 | 0.0 | 0.0

4. Primary Outcome: Number of Patients With Clinically Significant Changes to Vital Signs When Treated With EO-3021 as Monotherapy and in Combination With Ramucirumab or Dostarlimab
Time Frame: From the time of informed consent, for approximately 12 months (or earlier if the participant discontinues from the study), and through Safety Follow-up (28 days after the last dose
Measure: Count of Participants; unit: Participants
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0
Participants | 0.0 | 3.0 | 2.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Number of Patients With Clinically Significant Changes in Laboratory Tests When Treated With EO-3021 as Monotherapy and in Combination With Ramucirumab or Dostarlimab.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3.0 | 42.0 | 34.0 | 6.0 | 2.0 | 1.0
Participants | 0.0 | 3.0 | 2.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: The Estimate of Overall Response Rate (ORR) for the Efficacy Population.
Description: Tumor assessments were evaluated at baseline by computerized tomography (CT) or magnetic resonance imaging (MRI). The primary objective of this study was to determine the overall objective response rate (ORR) per investigator assessment, defined as confirmed complete response (CR; disappearance of all target lesions) + partial response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions) by RECIST v1.1.
Time Frame: Up to 24 months
Population: The Efficacy Evaluable Population includes all patients who receive at least one dose of EO-3021, have baseline measurable disease and at least one post baseline imaging assessment.
Measure: Count of Participants; unit: Participants
Groups:
- EO-3021 2.0 mg/kg in Combination With Dostarlimab: "In escalation, adult patients with advanced unresectable or metastatic gastric/GEJ adenocarcinoma will receive EO-3021 2.0 mg/kg in combination with dostarlimab every 3 weeks to determine MTD/RP2D(s).
  EO-3021: Anti-Claudin 18.2 antibody drug conjugate
  Dostarlimab: anti-PD-1 antibody"
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
Number analyzed (Participants) | 3 | 34 | 31 | 4 | 1 | 1
Participants | 1 | 5 | 4 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year 10 months
Arm/Group | EO-3021 Monotherapy 1.0 mg/kg | EO-3021 Monotherapy 2.0 mg/kg | EO-3021 Monotherapy 2.5 mg/kg | EO-3021 Monotherapy 2.9 mg/kg | EO-3021 2.0 mg/kg in Combination With Ramucirumab | EO-3021 2.0 mg/kg in Combination With Dostarlimab
All-Cause Mortality (participants affected / at risk) | 1/3 | 29/42 | 19/34 | 4/6 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 20/42 | 15/34 | 4/6 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 42/42 | 34/34 | 6/6 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EO-3021 Monotherapy 1.0 mg/kg (N=3) | EO-3021 Monotherapy 2.0 mg/kg (N=42) | EO-3021 Monotherapy 2.5 mg/kg (N=34) | EO-3021 Monotherapy 2.9 mg/kg (N=6) | EO-3021 2.0 mg/kg in Combination With Ramucirumab (N=2) | EO-3021 2.0 mg/kg in Combination With Dostarlimab (N=1)
Gastritis (Gastrointestinal disorders) | 0 | 4 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Upper Gasterointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary Tract Infection (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cerebral Infarction (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Impaired Gastric Temptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EO-3021 Monotherapy 1.0 mg/kg (N=3) | EO-3021 Monotherapy 2.0 mg/kg (N=42) | EO-3021 Monotherapy 2.5 mg/kg (N=34) | EO-3021 Monotherapy 2.9 mg/kg (N=6) | EO-3021 2.0 mg/kg in Combination With Ramucirumab (N=2) | EO-3021 2.0 mg/kg in Combination With Dostarlimab (N=1)
Nausea (Gastrointestinal disorders) | 2 | 25 | 20 | 5 | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 18 | 20 | 5 | 2 | 0
Fatigue (General disorders) | 1 | 18 | 9 | 3 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 14 | 10 | 2 | 1 | 0
Keratopathy (Eye disorders) | 1 | 11 | 13 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 8 | 6 | 3 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 7 | 6 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 5 | 6 | 2 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 8 | 5 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 6 | 3 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 5 | 5 | 1 | 0 | 1
Edema Peripheral (General disorders) | 1 | 3 | 5 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 8 | 1 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 3 | 4 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 2 | 5 | 0 | 0 | 1
Weight Decreased (Metabolism and nutrition disorders) | 0 | 5 | 2 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 4 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0 | 0 | 0
Hiccups (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 4 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 3 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 3 | 0 | 0 | 0
Malaise (General disorders) | 0 | 3 | 2 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 3 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT05980416/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT05980416/SAP_001.pdf